CLINICAL TRIAL: NCT06494917
Title: Investigation of the Effect of Manual Therapy and Pelvic Floor Exercises on Pelvic Floor Muscles in Women With Constipation
Brief Title: Investigation of the Effect of Manual Therapy and Pelvic Floor Exercises on Pelvic Floor Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Cihan Islek, master's degree student, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/02
Record Dates: First submitted 2024-06-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Colonic Inertia; Dyschezia; Constipation
Keywords: constipation; pelvic floor; manual therapy; exercise
MeSH Terms: conditions — Constipation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor exercises (Active Comparator): Diaphragmatic breathing training and Pelvic Floor Exercises will be applied.Participants will receive exercise training 5 days a week for 6 weeks.
  Interventions: Other: pelvic floor exercises
- Pelvic floor exercises and manual therapy techniques (Active Comparator): In addition to diaphragmatic breathing training and pelvic floor exercises, manual therapy methods will be applied. Participants will receive exercise training 5 days a week for 6 weeks. Manual therapy methods will be used 2 days a week for the first 2 weeks and then 1 day a week.
  Interventions: Other: Pelvic floor exercises and manual therapy techniques

INTERVENTIONS:
Other: pelvic floor exercises — First arm; Pelvic Floor Exercises (PFE) consisting of diaphragm breathing training, bridge exercise to strengthen the pelvic floor, 3-dimensional diaphragm exercise, 'I Love you massage' for intestinal motility, happy baby pose, child position exercise, full squat, adductor and iliopsoas stretching, mermaid position exercise, 'Shhh' sound exercise, 'Üüüü' sound exercise will be applied.
  Arms: pelvic floor exercises
Other: Pelvic floor exercises and manual therapy techniques — Second arm; Pelvic Floor Exercises (PFE) consisting of diaphragm breathing training, bridge exercise to strengthen the pelvic floor, 3-dimensional diaphragm exercise, 'I Love you massage' for intestinal motility, happy baby pose, child position exercise, full squat, adductor and iliopsoas stretching, mermaid position exercise, 'Shhh' sound exercise, 'Üüüü' sound exercise will be applied. In addition to diaphragmatic breathing training and pelvic floor exercises, manual therapy methods such as momentum minus mobilisation, sphincter opening, colon massage, global fascia manipulation, trigger point and myofascial release will be applied.
  Arms: Pelvic floor exercises and manual therapy techniques

SUMMARY:
The goal of this clinical trial is to Investigation of the effect of manual therapy and pelvic floor exercises on pelvic floor muscle in women with constipation. The main question[s] it aims to answer are:

* In addition to pelvic floor exercises, manual therapy applied to the pelvic floor muscles has no impact on constipation.
* In addition to pelvic floor exercises, manual therapy applied to the pelvic floor muscles has an impact on constipation.

Participants will apply pelvic floor exercises and manual therapy techniques. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

DETAILED DESCRIPTION:
* Female participants aged 18-55 years with constipation complaints will be recruited through social media and hospital outpatient clinics, and those who volunteer to participate will be enrolled in the study.
* Participants will be assessed as group 1 (pelvic floor exercises), group 2 (pelvic floor exercises + manual therapy techniques). Group 1 will receive diaphragmatic breathing training and then pelvic floor exercises to strengthen the pelvic floor.
* Group 2 will receive manual therapy methods consisting of Momentum Minus Mobilisation, Sphincter Opening, Colon Massage, Global Fascial Manipulation, Trigger Point and Myofascial Release in addition to Diaphragmatic Breathing Training and Pelvic Floor Exercises.
* Participants will receive exercise training 5 days a week for 6 weeks. Manual therapy methods will be used 2 days a week for the first 2 weeks and then 1 day a week. Initial assessment of participants and manual therapy applications will be done face to face. The exercises will be continued using the online telerehabilitation method.
* Both groups will be given nutritional advice, such as drinking plenty of water, eating fibre-rich foods and preferring foods that aid digestion. Participants will be advised to take their time every day, in the morning, at the same time, without rushing to defecate, preferring an squat toilet, which increases intra-abdominal pressure, half an hour after meals, but not for more than five minutes.If a European toilet is used, toilet training will be given about leaving a 15-18 cm long ridge under the feet.
* Both groups will be given assessment tests before and at the end of the trial and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Constipation in the last 6 months
* Being able to use smartphones and social media (whatsapp and instagram)
* Not having a health problem that prevents exercise
* Able to communicate
* Literate

Exclusion Criteria:

* Not had constipation in the last 6 months
* Pregnancy or recent pregnancy
* had surgery
* having a tumour
* Having vertigo Taking medication (use of bowel-regulating drugs)
* Previous physiotherapy for constipation problems
* Inflammatory bowel disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological female
Enrollment: 44 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Constipation Quality of Life questionnaire | will be evaluated at the first session and at the end of session 6
  evaluates constipation through daily individual health assessment and functioning. The highest score that can be obtained from the scale is 140 and the lowest score is 28. It is thought that quality of life is negatively affected as scores on the scale increase.

SECONDARY OUTCOMES:
Constipation Severity Scale | will be evaluated at the first session and at the end of session 6
  scale that is calculated as a sum of a 5-point ordinal frequency ratings for the six Rome III (IV) functional constipation questions. The lowest score is 0 and the highest is 73. A high score on the scale indicates that the symptoms are at a severe level.

OTHER OUTCOMES:
Bristol stool chart | will be evaluated at the first session and at the end of session 6
  Bristol stool chart is a medical aid designed to classify faeces into seven groups.
Rome IV Criteria | will be evaluated at the first session and at the end of session 6
  categorizes disorders of chronic constipation into four subtypes: (a) functional constipation, (b) irritable bowel syndrome with constipation, (c) opioid-induced constipation, and (d) functional defecation disorders, including inadequate defecatory propulsion and dyssynergic defecation
bowel diary | During the 6-week study
  a record you keep of when and how much faeces (poo) you passed or leaked during the day and overnight.

CONTACTS AND LOCATIONS:
Overall Officials: Serhad Bekir Sünbül, Study Chair — Cizre Dr. Selahattin Cizrelioğlu Devlet Hastanesi
Locations (1):
- Cizre Dr Selahattin Cizrelioglu State Hospital, Şırnak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SS, Bharucha AE, Chiarioni G, Felt-Bersma R, Knowles C, Malcolm A, Wald A. Functional Anorectal Disorders. Gastroenterology. 2016 Mar 25:S0016-5085(16)00175-X 10.1053/j.gastro.2016.02.009. doi: 10.1053/j.gastro.2016.02.009. Online ahead of print. PMID 27144630